CLINICAL TRIAL: NCT02987166
Title: A Pilot Study to Assess the Combination of High-Dose Conformal Radiation Therapy (HDCRT) and Pembrolizumab in Modulating Local and Systemic T-cell Responses in Advanced Malignancies
Brief Title: HDCRT Plus Pembrolizumab in Advanced Malignancies
Acronym: UVA-AM-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: James Larner, MD (Other)
Responsible Party: Sponsor-Investigator, James Larner, MD, James Larner, MD, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18488
Record Dates: First submitted 2016-11-30; First posted 2016-12-08 (Estimated); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Solid Tumor
Keywords: immunotherapy; pembrolizumab; MK-3475; High-dose conformal radiation therapy; HDCRT; advanced solid tumor
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: HDCRT administered with first dose of pembrolizumab (Experimental): Pembrolizumab (200 mg) plus HDCRT (24 Gy in 3 fractions of 8 Gy each for bone and/or soft tissue lesions; 30 Gy in 5 fractions of 6 Gy each for the prostate gland) are both administered beginning on day 1.
  Pembrolizumab (200 mg) will be administered on days 1, 43, 64, 85. Subjects who have measurable disease outside of the radiation field and who have derived benefit from the 4 doses of pembrolizumab may continue to receive pembrolizumab every 3 weeks for up to 2 years.
  HDCRT will be administered to the primary tumor and/or sites of metastatic disease (1 or more sites permitted) over a period of 3-5 days. The length of time for administration of the HDCRT will depend on the site of disease that is to be radiated. HDCRT will begin on day 1.
  Interventions: Radiation: High-Dose Conformal Radiation Therapy; Drug: Pembrolizumab
- Arm B: HDCRT administered between doses 1& 2 of pembrolizumab (Experimental): Pembrolizumab (200 mg) begins on day 1. HDCRT (24 Gy in 3 fractions of 8 Gy each for bone and/or soft tissue lesions; 30 Gy in 5 fractions of 6 Gy each for the prostate gland) begins on day 22.
  Pembrolizumab (200 mg) will be administered on days 1, 43, 64, 85. Subjects who have measurable disease outside of the radiation field and who have derived benefit from the 4 doses of pembrolizumab may continue to receive pembrolizumab every 3 weeks for up to 2 years.
  HDCRT will be administered to the primary tumor and/or sites of metastatic disease (1 or more sites permitted) over a period of 3-5 days. The length of time for administration of the HDCRT will depend on the site of disease that is to be radiated. HDCRT will begin on day 22.
  Interventions: Radiation: High-Dose Conformal Radiation Therapy; Drug: Pembrolizumab
- Arm C: HDCRT administered prior to first dose of pembrolizumab (Experimental): Pembrolizumab (200 mg) begins on day 1. HDCRT (24 Gy in 3 fractions of 8 Gy each for bone and/or soft tissue lesions; 30 Gy in 5 fractions of 6 Gy each for the prostate gland) begins on day 1.
  Pembrolizumab will be administered on days 22, 43, 64, and 85. Subjects who have measurable disease outside of the radiation field and who have derived benefit from the four doses of pembrolizumab may continue to receive pembrolizumab every 3 weeks for up to 2 years.
  HDCRT will be administered to the primary tumor and/or sites of metastatic disease (1 or more sites permitted) over a period of 3-5 days. The length of time for administration of the HDCRT will depend on the site of disease that is to be radiated. HDCRT will begin on day 1.
  Interventions: Radiation: High-Dose Conformal Radiation Therapy; Drug: Pembrolizumab

INTERVENTIONS:
Radiation: High-Dose Conformal Radiation Therapy — 24 Gy in 3 fractions of 8Gy each for bone and/or soft tissue lesions
  30 Gy in 5 fractions of 6 Gy each for prostate gland
  Other Names: HDCRT
Drug: Pembrolizumab — 200 mg
  Other Names: Keytruda; MK-3475

SUMMARY:
This study is a pilot study to evaluate high-dose conformal radiation therapy (HDCRT) administered in combination with pembrolizumab in patients with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a histologically or cytologically proven advanced solid tumor malignancy for which palliative radiation is recommended. In solid tumors where pembrolizumab has been approved for use, patients may receive pembrolizumab as indicated, in the context of this protocol. In solid tumors where pembrolizumab has not been approved for use, the following criteria apply:

  * Patients must be resistant to at least 1 prior conventional chemotherapy regimen or other standard of care regimen,
  * Patient must have no remaining conventional treatment options proven to provide long-term disease control, and
  * Patient has declined other conventional treatment options
* Palliative radiation therapy may be recommended for primary tumor and/or any metastatic site that is accessible to biopsy.
* At least one site of disease that is accessible to radiation and multiple biopsies. Subjects may have disease that is encompassed within the radiation field or may have known disease both inside and outside of the radiation field.
* Must be able to provide tissue from 2-3 separate biopsy procedures that will be completed throughout the course of the study.
* A performance status of 0, 1 or 2 on the ECOG Performance Scale.
* Subjects must demonstrate adequate organ function.
* A life expectancy ≥ 6 months.

Exclusion Criteria:

* Requires urgent treatment with cytotoxic chemotherapy or other therapy is indicated.
* A diagnosis of immunodeficiency.
* A known history of active TB (Bacillus Tuberculosis).
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with untreated brain metastases and patients who have had brain metastases re-treated with radiation will be excluded. Patients whom have either midline shift, or any signs of herniation (even if disease has been treated with GK) will be excluded. Subjects with previously treated brain metastases may participate provided they are 1) stable (without clinical evidence of progression) 2) are out at least 10 days from CNS radiation and 3) and are not using steroids as part of treatment for their brain lesions for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Active autoimmune disease that has required systemic treatment in the past 2 years.
* A history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* An infection requiring systemic therapy.
* Pregnancy.
* HIV positivity.
* Evidence of active Hepatitis B virus or Hepatitis C virus.
* Significant cardiovascular disease including unstable angina pectoris, uncontrolled hypertension, uncontrolled arrhythmias, or severe valvular heart disease, or a myocardial infarction within 6 months prior to the first dose of study treatment.
* Active bleeding disorders or evidence of chronic or acute disseminated intravascular coagulation (DIC).
* Class III or IV heart disease (New York Heart Association classification).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Safety: adverse event profile | 30 days post-treatment for adverse events; 90 days post-treatment for serious adverse events
  Obtain preliminary data on the safety of HDCRT with immunotherapy, delivered concurrently (Arm A) or sequentially (Arms B and C)
Immunologic: effect on T cell tumor infiltration | through day 43
  Estimate the effect of HDCRT, pembrolizumab, and the combination of HDCRT and pembrolizumab on CD8+ T cell and CD4+ T regulatory cell infiltration in tumors.

SECONDARY OUTCOMES:
Immunologic: effect on lymphocyte composition of blood | up to year 2
  Estimate the effect of HDCRT, pembrolizumab, and the combination of HDCRT and pembrolizumab on the lymphocyte composition of blood over time.

CONTACTS AND LOCATIONS:
Overall Officials: James Larner, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No